CLINICAL TRIAL: NCT00870402
Title: Effect of Aldosterone Antagonism in the Reduction of Albuminuria and Diastolic Disfunction of Patients With Diabetic Nephropathy.
Brief Title: Aldosterone in Diabetic Nephropathy
Acronym: ALDODN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Francisco Espinoza Villegas, Departament of Internal Medicine, University of los Andes
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA08I20032
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Diabetic Nephropathy
Keywords: aldosterone; albuminuria; diastolic disfunction; hyperkalemia
MeSH Terms: conditions — Diabetic Nephropathies; Albuminuria; Hyperkalemia | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Spironolactone
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — 25 mg per day for 9 months
  Arms: 1
Drug: Placebo — Placebo 1 tablet per day for nine months
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether spironolactone are effective in the reduction of albuminuria and diastolic disfunction of subjects with diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic subjects with maximum ten years after diagnostic
* Diabetic nephropathy with albuminuria
* Normal renal function
* Diastolic disfunction
* Taking a IECA or ARA drug family previously

Exclusion Criteria:

* Diabetics subjects with macroangiopathy
* Acute coronary syndrome in the three months before
* Hyperkalemia > 5.5 mEq/L
* Pregnancy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Reduction of albuminuria | 9 months

SECONDARY OUTCOMES:
Reduction of diastolic disfunction | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Los Andes, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Kozie DW, Hassul M, Kimm J. Effect of tympanic membrane perforations on air caloric response in monkeys. Trans Sect Otolaryngol Am Acad Ophthalmol Otolaryngol. 1976 Mar-Apr;82(2):203-9. No abstract available. PMID 820032
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592